CLINICAL TRIAL: NCT00352521
Title: Dynamic Contrast-Enhanced Magnetic Resonance Imaging With Bevacizumab in Combination With Irinotecan for Malignant Gliomas
Brief Title: Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI) With Bevacizumab and Irinotecan for Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00012387; DUMC-8053-05-12R0; CDR0000481476 (Other: NCI)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma; recurrent adult brain tumor; adult glioblastoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult pineal gland astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Glioma; Glioblastoma; Gliosarcoma; Brain Neoplasms; Ependymoma; Oligodendroglioma | interventions — Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab and irinotecan (Experimental): The bevacizumab will be dosed at 10 mg/kg every 14 days (days 1, 15 and 29) and the irinotecan on days 2, 15, and 29 of the first six week schedule. The irinotecan dose will depend on whether the patient is on an enzyme-inducing antiepileptic drug (EIAED). If the patient is on an EIAED, the patient will receive 340 mg/m2 on days 2, 15, and 29 of the first six week schedule. If the patient is not on an EIAED, the dose of irinotecan will be 125 mg/m2 on days 2, 15, and 29 of the first six week schedule. After the first cycle, the irinotecan and bevacizumab will be given on days 1, 15 and 29.
  Interventions: Drug: bevacizumab; Drug: irinotecan; Procedure: dynamic contrast-enhanced magnetic resonance imaging

INTERVENTIONS:
Drug: bevacizumab
  Other Names: Avastin
Drug: irinotecan
  Other Names: Camptosar
Procedure: dynamic contrast-enhanced magnetic resonance imaging

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also block blood flow to the tumor. Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with irinotecan may kill more tumor cells. Diagnostic procedures, such as MRI, may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with irinotecan works in treating patients with recurrent malignant glioma and how well MRI predicts response to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Examine the effect of bevacizumab and irinotecan on vascular permeability and blood flow in patients with recurrent malignant gliomas.

Secondary

* Determine the reproducibility of dynamic contrast-enhanced (DCE-MRI) in malignant gliomas.
* Determine the predictive value of DCE-MRI in patients with recurrent malignant gliomas treated with bevacizumab and irinotecan.
* Describe the activity of the combination of bevacizumab with irinotecan as measured by response rate and progression-free survival.
* Describe the toxicity associated with the administration of bevacizumab with irinotecan.

OUTLINE: Patients receive bevacizumab IV on days 1, 15, and 29 and irinotecan IV on days 2, 15, and 29 during the first 6-week cycle. After the first cycle, the irinotecan and bevacizumab will be given on days 1, 15 and 29. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

Patients also undergo dynamic contrast-enhanced MRI 4 times.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of any of the following malignant gliomas:

  * Glioblastoma multiforme
  * Anaplastic astrocytoma
  * Grade 3 or greater WHO astrocytic, oligodendroglial, or mixed glial tumors that were initially diagnosed by histologic examination of a tumor specimen obtained from biopsy or resection
* Recurrent disease

  * No more than 3 prior recurrences
* Measurable recurrent or residual primary CNS neoplasm on contrast-enhanced MRI or CT scan
* No evidence of CNS hemorrhage on baseline MRI or CT scan

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Hematocrit > 29%
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 125,000/mm³
* Creatinine < 1.5 mg/dL
* SGOT < 1.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active infection
* No significant traumatic injury within the past 28 days

PRIOR CONCURRENT THERAPY:

* At least 6 weeks since prior surgical resection
* More than 28 days since prior major surgical procedure or open biopsy
* More than 7 days since prior minor surgical procedure, fine-needle aspirations, or core biopsies
* At least 6 weeks since prior chemotherapy*
* At least 4 weeks since prior radiotherapy*
* No concurrent immunosuppressive agents
* No concurrent therapeutic anticoagulation
* Concurrent corticosteroids allowed if dose has been stable for 1 week prior to study entry NOTE: * Unless there is unequivocal evidence of progressive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Correlation of the acute permeability and blood flow response (24-48 hours) with progression-free survival (PFS) | 1 year
  Assessed by DCE-MRI

SECONDARY OUTCOMES:
Overall Survival and Tumor Response | 2 years
Incidence and severity of central nervous system (CNS) hemorrhage and systemic hemorrhage | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James J. Vredenburgh, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States